CLINICAL TRIAL: NCT00586534
Title: Developing Computer Based Treatments for Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00011048; R01DA026454 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Cocaine Addiction
Keywords: crack, cocaine, addiction treatment, virtual reality
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I/GDC (Active Comparator): NIDA approved Individual/Group Drug Counseling (I/GDC) cocaine treatment
  Interventions: Behavioral: I/GDC
- I/GDC + VR/CER (Experimental): Second Arm:NIDA approved Individual/Group Drug Counseling (I/GDC) cocaine treatment plus virtual reality (VR) based cue exposure/extinction software and cellular phone-based computerized extinction reminder (CER) technology for use in high-risk situations outside treatment sessions.
  Interventions: Behavioral: I/GDC + VR/CER

INTERVENTIONS:
Behavioral: I/GDC + VR/CER — NIDA approved Individual/Group Drug Counseling (I/GDC) cocaine treatment plus virtual reality (VR) based cue exposure/extinction software and cellular phone-based computerized extinction reminder (CER) technology for use in high-risk situations outside treatment sessions.
  Other Names: drug counseling; group drug counseling; individual drug counseling; virtual reality; exposure/extinction software; cellular phone based computerized extinction reminder
  Arms: I/GDC + VR/CER
Behavioral: I/GDC — NIDA approved Individual/Group Drug Counseling (I/GDC) cocaine treatment
  Other Names: drug counseling; group drug counseling; individual drug counseling
  Arms: I/GDC

SUMMARY:
The purpose of our research is to examine the promise of a new computer based approach to use in usual drug counseling when treating crack cocaine addiction.

DETAILED DESCRIPTION:
This is the next part of the project under a National Institute of Drug Abuse-funded R01 treatment development study with the purpose of developing a computer-based augmentation of standard drug counseling for cocaine dependence. This project has received additional funding from NIDA. Specifically, the aims of the next part of the proposal are to develop and manualize a cue-exposure based cocaine treatment using virtual reality (VR) based cue exposure/extinction software and cellular phone-based computerized extinction reminder (CER) technology for use in high-risk situations outside treatment sessions. We will enroll a total of 270 cocaine dependent subjects in order to meet the target goal of 180 subjects in treatment. This randomized clinical trial will be conducted in order to determine the acceptability and feasibility of this treatment to subjects and therapists, and to obtain treatment outcome effect size estimates. Specifically, during the next stage of the study, 180 cocaine dependent individuals will be randomly assigned to receive a NIDA approved Individual/Group Drug Counseling (I/GDC) cocaine treatment or I/GDC plus VR/CER. Matching between treatment groups will be based on age, sex, severity of crack use (using the Addiction Severity Index), and presence or absence of antisocial personality disorder. Treatment assignment will be conducted using a computerized urn matching program by the off-site study statistician. Current psychiatric diagnoses will be assessed, as will changes in crack use. Comprehensive assessments will be conducted during treatment at baseline, and at a six-month and twelve-month follow-up. To measure outcomes, substance use will be assessed via self-report and urinary analysis three times weekly during 24 weeks of active treatment and weekly during six month and twelve month of follow-up assessment.

This new larger part of project follows work we have conducted in a NIDA-funded pilot project over the past four years, developing the complementary intervention. In our preliminary studies (Phase I a/b), we conducted focus groups, an open trial, and a small randomized controlled trial (n = 53) to demonstrate the promise of the novel intervention. The pilot phase I a/b portion enrolled 171 subjects (signed consent) at Duke. 19 of 53 completed the treatment portion. During Phase 1a, the VR and CER technology was developed and refined using two small open clinical trials. At the conclusion of Phase 1a, a treatment manual detailing the rationale and parameters of VR and CER technology was completed. Next, as mentioned, a Phase Ib pilot randomized clinical trial was conducted in order to determine the acceptability and feasibility of this treatment to patients and therapists, and to obtain treatment outcome effect size estimates.

ELIGIBILITY:
Inclusion Criteria:

* Meets SCID-I criteria for cocaine dependence; crack cocaine is primary substance of abuse
* Consents to outpatient treatment for drug addiction
* Resides within commuting distance of treatment

Exclusion Criteria:

* Full criteria met for psychotic disorders
* Full criteria met for current mania
* IQ less than 70
* Unable to give consent
* Can not read
* Current and chronic absence of shelter
* Impending jail/prison for more than three weeks (problems which by their presence or severity preclude ability to attend or understand treatment and/or requires priority treatment over substance use treatment)
* Court order to treatment or to jail, or agency order to treatment or loss of child custody (due to inability to freely drop-out of treatment)
* Refuses to discontinue current drug abuse treatment or refuses random assignment
* If the potential participant lives with or is in an intimate relationship with another participant currently being treated in the study, they will be told that they cannot participate until that housemate or partner has completed treatment in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2007-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Urinalyses | 1 year
  urinary analysis will be conducted three times weekly during 24 weeks of active treatment. During the booster phase (months 7-9), UA's will occur once monthly, before the booster sessions and again at 12 months. Urine will be tested for cocaine, marijuana, opiates, amphetamines, and benzodiazepines

SECONDARY OUTCOMES:
Physiological measures: skin conductance, heart rate, and skin temperature | Intake, 6 month, 9 month, and 12 month follow-up assessments
  They will be measured using Ag-AgCl electrodes. They will be measured during a 5 minute videotape showing cocaine paraphernalia and use.
Interview measures: Structured Clinical Interview for DSM-IV, Axis I (SCID-I), Addiction Severity Index | Intake, 6 month, 9 month, and 12 month assessments.
Self-report measures of Substance use [e.g., TLFB; Minnesota Cocaine Craving Questionnaire (MCCS); Cocaine Craving Questionnaire (CCQ)] | Intake assessment, 6 months, 9months, 12 months
HIV Risk Behaviors | 6 months, 9 months, 12 months
  The 11-item HIV Risk Behavior Scale (a brief self-report measure using a 6-point Likert-type scale, will be utilized at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Rosenthal, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States